CLINICAL TRIAL: NCT07109713
Title: A Randomized, Parallel, Controlled Trial Investigating the Effects a Cranberry-Based Products on the Female Microbiome
Brief Title: The Effect Cranberry-Based Products on the Female Microbiome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ocean Spray Cranberries, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Bio-2502
Record Dates: First submitted 2025-07-31; First posted 2025-08-07 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Vaginal Microbiome; Gut Microbiome; Gut Health
Keywords: vaginal microbiome; gut microbiome; cranberry; polyphenols
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cranberry beverage (Active Comparator): Participant will receive 8 oz of cranberry beverage to consume each day
  Interventions: Dietary Supplement: Active
- Placebo Beverage (Placebo Comparator): Participant will receive 8 oz of placebo beverage to consume each day
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Active — Cranberry Beverage
  Arms: Cranberry beverage
Dietary Supplement: Placebo — Placebo Beverage
  Arms: Placebo Beverage

SUMMARY:
The overall objective of this clinical trial is to compare the effects of a cranberry-based product to a placebo-control product on vaginal and GI microbiome outcomes and associated participant reported outcomes in generally healthy pre-menopausal women

DETAILED DESCRIPTION:
Among various strategies explored to modulate the composition and function of different microbiomes, dietary interventions, like the consumption of cranberry-based products have garnered interest due to their historical use and emerging scientific evidence suggesting beneficial effects on host health. Cranberries are rich in bioactive compounds, notably polyphenols such as proanthocyanidins, which have been investigated for their potential to influence microbial adhesion and growth, especially in the genitourinary tract. While cranberry phenolic compounds generally exhibit poor bioavailability, they have been shown to be metabolized by gut microbiota through fermentation in the distal intestine, yielding bioavailable and bioactive bacteria-derived metabolites. These findings highlight the critical need to understand the potential crosstalk between human microbiome ecosystems and how dietary cranberries might modulate this interaction to impact health outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Pre-menopausal female,
* 18 - 45 years of age (inclusive) at visit 1.
* History of regular menstrual cycles (21-35 d per cycle or at the investigator's discretion) for at least 3 months prior to visit 1. Participants that are using contraceptives (IUD, patch, or pills) must be on a stable dose, defined as no change in medication regimen, within 90 days of visit 1 (or within 6 months of visit 1 for copper IUD users) and no plans to change hormonal contraceptive use during the study.
* BMI ≥18.5 to <30.0 kg/m2 at visit 1.
* Willing to adhere to all study procedures, including lifestyle considerations (see section 6.2), and sign forms providing informed consent to participate in the study and authorization to release relevant protected health information to the Clinical Investigator.

Exclusion Criteria:

Women's health related criteria

•Female who is pregnant, planning to be pregnant during the study period, lactating, or is of childbearing potential and is unwilling to commit to the use of a medically approved form of contraception throughout the study period.

General health related criteria

* Participant has a history or presence of any gastrointestinal condition that could potentially interfere with absorption of the study product (e.g., inflammatory bowel syndrome, celiac disease, history of gastric bypass surgery).
* History or presence of clinically important cardiac, renal, hepatic, endocrine (including diabetes mellitus), pulmonary, gastrointestinal, biliary, pancreatic, or neurological disorders that may affect the participant's ability to adhere to the study protocol and/or affect study outcomes, in the judgment of the Investigator.
* Uncontrolled hypertension (systolic blood pressure ≥140 mm Hg or diastolic blood pressure ≥90 mm Hg) as defined by the blood pressure measured at visit •Stable use of hypertension medication is allowed (defined as no change in medication regimen ≤ 90 d of visit 1).
* Any signs or symptoms of active infection of clinical relevance (e.g., urinary tract or respiratory) within 5 days prior to any test visit. If an infection occurs during the study period, test visits should be rescheduled until all signs and symptoms have resolved and any treatment has been completed at least 5 days prior to testing.
* History or presence of cancer in the prior 2 years, except for non-melanoma skin cancer.
* History of any major trauma or major surgical event within 2 months of visit 1.
* Subject has elective hospitalizations planned (e.g., elective cosmetic procedures) during the study period.
* Underwent an endoscopy or colonoscopy preparation within 3 months prior to visit 1.

Exclusionary products related criteria

* Recent history of (within 12 months of screening; visit 1) or strong potential for alcohol or substance abuse. Alcohol abuse is defined as >14 drinks per week (1 drink = 12 oz beer, 5 oz wine, or 1½ oz distilled spirits).
* Use of tobacco/nicotine products (e.g., cigarette smoking, vaping, chewing tobacco) within 12 months of visit 1.
* Habitual users (i.e., daily or almost daily) of marijuana and hemp products, including CBD products, and willing to abstain from use throughout the study period (topical creams/lotions are allowed). Occasional use (e.g., couple times a month) within 12 months of visit 1 is allowed but requires at least a 14 d washout prior to visit 1 and the participant must be willing to refrain from use during the study.
* Unstable use of any prescription medication, where stable use is defined as no change in dose or medication type within 90 days of visit 1. This exclusion criterion does not include hormonal contraceptives.
* Exposed to any non-registered drug product within 30 days prior to visit 1.
* Antibiotic use within 30 d of visit 1 and throughout the study period.
* Steroid use within 30 d of visit 1 and throughout the study period.
* Current habitual user (≥ 3 days/week ≤ 1 month of visit 1) of anti-inflammatory medications (e.g., NSAIDs, acetaminophen, etc.).
* Use of medications (over-the-counter or prescription) and/or dietary supplements, known to influence GI function, including but not limited to, pre-, post-, and probiotic supplements, fiber supplements, laxatives, enemas, suppositories, H2 blockers, proton pump inhibitors, antacids, anti-diarrheal agents, anti-depressants, and/or anti-spasmodic within 30 d of visit 1 and throughout the study period. Standard multivitamin and mineral supplements are allowed.
* Willing to avoid consuming probiotics or fermented foods within 14 d of visit 1 and throughout the study period.
* Willing to avoid consuming high-polyphenol foods and supplements [e.g., dark colored and polyphenol-rich fruits (berries, grapes, pomegranates, cherries, grapefruit, black currant, plum) and their processed food/juice and related supplement products (e.g. grape seed extract, green tea extract); red wine; dark chocolate; cranberry extract supplements] throughout the study period.

General safety related criteria

* Known sensitivity, intolerability, or allergy to any of the study products or their excipients.
* Any condition the Investigator believes would interfere with the participant's ability to provide informed consent or comply with the study protocol, which might confound the interpretation of the study results or put the person at undue risk

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08-05 (Actual); Primary Completion 2025-12-19 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
Vaginal Microbiome | 4 weeks
  The number of participants exhibiting a Lactobacillus-dominant CST vaginal microbiome following the 28-day intervention

SECONDARY OUTCOMES:
Vaginal Microbiome Diversity | 4 weeks
  Microbiome diversity (e.g., α-diversity, β-diversity, Bray-Curtis dissimilarity, relative change in taxa abundance)
Vaginal pH | 4 weeks
  vaginal pH
GI microbiome | 4 weeks
  Microbiome diversity (e.g., α-diversity, β-diversity, Bray-Curtis dissimilarity, relative change in taxa abundance)
Vaginal health questionairre | 4 weeks
  Vaginal health visual analog score: itching, dryness, discharge, odor. This is a scale from 0-3 with 3 being the most bothersome score
Gastrointestinal Symptom Rating Scale (GSRS) | 4 weeks
  GI symptoms are measured using a Gastrointestinal Symptom Rating Scale (GSRS), which ranges from 1 to 7 per item, with higher scores indicating worse gastrointestinal symptoms
RAND SF-36 component scores | 4 weeks
  To assess overall physical and mental health-related quality of life, scores were reported using the RAND 36-Item Health Survey (SF-36), with Physical and Mental Component Summary scores ranging from 0 to 100, where higher scores indicate better health status
Bristol Stool Scale score | 4 weeks
  Stool consistency was measured using the Bristol Stool Form Scale (BSFS), which categorizes stool into seven types ranging from 1 (hard, indicative of constipation) to 7 (liquid, indicative of diarrhea), with types 3 and 4 considered most typical of healthy bowel movements

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Antoo, MD, Principal Investigator — BioFortis
Locations (1):
- Biofortis, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No